CLINICAL TRIAL: NCT06706063
Title: Clinical and Ultrasonographic Evaluation of Spasticity in Hemiplegic Patients
Brief Title: Ultrasonograpy in Hemiplegic Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, Ass. Prof., Afyonkarahisar Health Sciences University
Other Study IDs: SAUSG
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Hemiplegia; Hemiparesis After Stroke; Spasticity
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Ultrasonography of muscles — The biceps brachii, flexor digitorum superficialis and profundus muscles and gastrocnemius muscles of the participants on the affected and unaffected sides will be evaluated ultrasonographically. Two researchers (with at least 5 years of experience in ultrasound imaging) blinded to the clinical evaluations of the patients and previous measurements will evaluate the same patients at two different times to test interobserver reproducibility. Muscle thickness, fascicle length and pennation angle will be recorded on B-mode imaging. In addition, elastographic evaluation will be performed on the same muscles and strain rate will be recorded.

SUMMARY:
The aim of this study was to evaluate the architectural changes and muscle stiffness of the upper and lower extremity muscles in our hemiplegic patients ultrasonographically and to investigate their relationship with clinical assessment scales.

DETAILED DESCRIPTION:
Spasticity has been defined as "disorganized sensorimotor control resulting from upper motor neuron lesion, manifested as intermittent or continuous involuntary activation of muscles". Its high prevalence and limited effectiveness of current treatment options make spasticity an important health problem in neurological rehabilitation.

The commonly used tools for the assessment of spasticity are subjective clinical scales, including the Ashworth Scale (AS), Modified AS (MAS), Tardieu Scale (TS), Modified TS (MTS), and Tone Assessment Scale (TAS). Most of these scales have limitations regarding reliability and inter-examiner reproducibility. Many uncontrollable or unstable factors can affect the measurement results.

On the other hand, spasticity can be assessed objectively using isokinetic dynamometers or electromyography (EMG). However, EMG data can be affected by various factors (electrode placement, muscle atrophy, skin resistance, etc.). These quantitative and objective methods require technological skills and equipment and can only assess a limited number of muscles. Ultrasonography has been used to determine muscle size (muscle length and volume), architectural features (thickness, cross-sectional area, fascicle length, and pennation angle), as well as content features (e.g., stiffness) of spastic muscles in patients with central nervous system injuries. In clinical practice, muscle atrophy-loss of contractile tissue-is usually measured by cross-sectional area or thickness (reflecting cross-sectional area) in spastic patients. Ultrasound is also useful for measuring fascicle length and pennation angle, architectural features that determine the muscle movement and force generated along the line of tension, respectively. The fascicle length of the affected muscle on the hemiparetic side of stroke patients was found to be shorter than in nonparetic and healthy controls. In addition to architectural changes, excessive stiffness felt during movement of the segments around the joint causes movement impairment in patients with spasticity. Ultrasound elastography has recently enabled physicians to accurately measure passive muscle stiffness. It has been found that spastic muscle stiffness increases in patients with central nervous system injuries.

Muscles frequently evaluated by ultrasound elastography are biceps and gastrocnemius muscles, which are reported to be highly affected by spasticity. However, the lack of a standard measurement protocol and the variability of elasticity in patients need to be addressed. Since there are few studies investigating the application of ultrasound elastography techniques for measuring muscle stiffness, future studies are needed to understand the mechanical properties of the muscles and to obtain a standard and reliable protocol. In the literature, only one study has evaluated forearm muscles elastographically and found that the elasticity ratio was lower on the hemiplegic side compared to the non-hemiplegic side.

The aim of this study was to evaluate the architectural changes and muscle stiffness of the upper and lower extremity muscles in our hemiplegic patients ultrasonographically and to investigate their relationship with clinical assessment scales.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70
* Unilateral hemiplegia
* At least 3 months since cerebrovascular accident

Exclusion Criteria:

* Operation or fracture in the last 3 months
* Botulinum toxin injection in the last 6 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 hemiplegic patients aged between 40-70 years, with unilateral hemiplegia, and at least 3 months after a cerebrovascular accident, who applied to the AFSU Department of Physical Medicine and Rehabilitation will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Spasticity Evaluation | T0 (First day), T1 (Second day)
  Spasticity was planned to be evaluated with the Modified Ashworth Scale (MAS). In the MAS, patients are evaluated out of 5 points. 0 indicates no increase in muscle tone, and 4 indicates that the extremity is rigid in the flexion and extension directions.
Fugl Meyer Assessment Questionnaire | T0 (First day), T1 (Second day)
  Fugl-Meyer Motor Assessment Scale was developed to quantitatively assess sensorimotor recovery after stroke. It was prepared based on Brunnstrom's motor recovery stages. Validity and reliability study was conducted in Turkish. The total score is between 0-66 and higher scores indicates better motor functions.
Neurophysiological Evaluation | T0 (First day), T1 (Second day)
  Brunnstrom Staging is a test that evaluates the motor development of hemiplegic patients. In this test, the neurophysiological recovery process of the hemiplegic patient is defined as 6 stages. According to this staging, the lowest stage is stage 1 (flaccid, no voluntary movement stage), and the highest stage is stage 6 (isolated joint movement stage). In Brunnstrom staging, the hand, upper extremity and lower extremity are evaluated separately.
Ultrasonographic Evaluation | T0 (First day), T1 (Second day)
  The biceps brachii, flexor digitorum superficialis and profundus muscles and gastrocnemius muscles of the participants on the affected and unaffected sides will be evaluated ultrasonographically. Two researchers (with at least 5 years of experience in ultrasound imaging) blinded to the clinical evaluations of the patients and previous measurements will evaluate the same patients at two different times to test interobserver reproducibility. Muscle thickness, fascicle length and pennation angle will be recorded in B-mode imaging. In addition, elastographic evaluation will be performed on the same muscles.

SECONDARY OUTCOMES:
Functional Independence Measurement (FIM) | T0 (First day), T1 (Second day)
  It is a scale that evaluates the performance of individuals regarding daily living activities. It consists of 18 items and evaluates the functions of individuals in 2 main sections: physical/motor function (13 items) and cognitive function (5 items). The items are also grouped under 6 subheadings (self-care, sphincter control, transfers, movement, communication and social perception). Each item is scored between 1-7; 1 indicates full assistance and 7 indicates full independence. The total score varies between 18-126 (full dependency-full independence). Adaptation, validity and reliability studies of the scale to the Turkish population have been conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University Health Application and Research Center Physical Medicine and Rehabilitation Clinic, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No